CLINICAL TRIAL: NCT02848859
Title: Improving Sleep for Healthy Hearts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Susan Redline, Senior Physician, Division of Sleep and Circadian Disorders, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000845
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Insomnia; Coronary Heart Disease
Keywords: cognitive behavioral therapy for insomnia; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: Go! to Sleep (Active Comparator): We are using a web-based cognitive behavioral therapy program called Go! to Sleep. Go! to Sleep is an interactive online program developed by specialists in Cleveland Clinic's Wellness Institute and Sleep Disorders Center. The program is a 6 week self-help program that uses cognitive behavioral therapy techniques that have been proven to be effective in decreasing symptoms of insomnia.
  Interventions: Behavioral: Go! to Sleep; Behavioral: General Sleep Education
- General Sleep Hygiene Education (Placebo Comparator): General Sleep Hygiene Education is the first step in the treatment of any sleep disorder. Both arms will have access to a Harvard sleep education web site that provides general information about sleep as well as sleep hygiene.
  Interventions: Behavioral: General Sleep Education

INTERVENTIONS:
Behavioral: Go! to Sleep — This is an online interactive program that delivers cognitive behavioral therapy for insomnia via the internet.
  Other Names: web-based cognitive behavioral therapy
  Arms: Intervention: Go! to Sleep
Behavioral: General Sleep Education — Providing patients information on healthy sleep and habits to promote healthy sleep.

SUMMARY:
This is a pilot study randomizing patients with insomnia and coronary heart disease to either general sleep hygiene counseling and web-based cognitive behavioral therapy for insomnia versus general sleep hygiene counseling alone (followed by the cognitive behavioral therapy at a later date).

DETAILED DESCRIPTION:
For this pilot study, the investigators will recruit up to 30 participants with insomnia and coronary heart disease. Another 30 patients will be recruited from another institution. Patients will be screened with a modified version of the Insomnia Severity Index (ISI), a brief self-report instrument validated for identifying insomnia. The investigators will modify the ISI to include exclusionary criteria. The investigators will randomize participants to 6 weeks of access to web based cognitive behavioral therapy for insomnia (wCBT-I) using an internet based CBT-I program plus education provided through access to the Harvard Sleep Education web site (which provides general sleep education information only) compared to 6 weeks of access to the Harvard Sleep Education web site, followed by access to the web-CBT program (a wait list control group). The investigators will test the hypothesis that use of wCBT-I improves sleep quality and sleep duration as measured by sleep diaries and the ISI. A secondary goal of the study is to assess the recruitment yields, retention and adherence rates.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for at least mild insomnia based on the Insomnia Severity Index questionnaire results
* have established coronary disease defined by: a) prior myocardial infarction or a coronary artery revascularization procedure; b) angiographically documented stenosis (>70%) of a major coronary artery; or c) prior ischemic stroke without major functional impairment.
* minimum age of 18 years old.

Exclusion Criteria:

* no daily access to a computer with an internet connection
* visual impairment preventing use of a computer
* inability to read English
* severe uncontrolled medical or psychiatric problems
* heart failure with reduced ejection fraction <35%
* high depressive symptoms (PHQ > 15)
* drowsy driving
* >3 days per week use of hypnotic medications
* known untreated sleep disordered breathing, narcolepsy, or restless leg syndrome
* shift-workers
* prior exposure to CBT-I treatment
* dialysis patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Insomnia Severity Index score at 6 weeks | At baseline, at 6 weeks, and in the treatment arm at 12 weeks.
  It is a 7 item, validated questionnaire to determine severity of insomnia symptoms.

SECONDARY OUTCOMES:
Change in sleep duration from baseline to 6 weeks | At baseline, at 6 weeks, and in the treatment arm at 12 weeks.
  The investigators will use sleep diaries that participants fill out for 1 week at baseline and at 6 weeks to compare sleep duration between arms as well as at 12 weeks in the treatment arm only to assess duration of treatment effect.
Change in mood assessed using the Patient Health Questionnaire-8 from baseline to 6 weeks | At baseline, at 6 weeks, and in the treatment arm at 12 weeks.
  The investigators will use the Patient Health Questionnaire-8 to measure depressive symptoms
Change in sleepiness assessed using the Epworth Sleepiness Questionnaire from baseline to 6 weeks | At baseline, at 6 weeks, and in the treatment arm at 12 weeks.
  The investigators will use the Epworth Sleepiness questionnaire to measure sleepiness.
Change in blood pressure from baseline to 6 weeks | At baseline and at 6 weeks
  The investigators will measure seated blood pressure in triplicate and use the average of the latter two readings for blood pressure (taken at baseline and 6 week visits).
Change in heart rate from baseline to 6 weeks | At baseline and at 6 weeks
  The investigators will measure seated heart rate in triplicate and use the average of the latter two readings for heart rate(taken at baseline and 6 week visits).
Change in Quality of life at baseline and 6 weeks | At baseline, at 6 weeks, and in the treatment arm at 12 weeks.
  The investigators will measure this using the Duke Health Profile, another validated questionnaire to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Sogol Javaheri, MD, MA, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States